CLINICAL TRIAL: NCT06587386
Title: The Minimum Effective Dose (ED90) of Liposomal Bupivacaine for Preserving Motor Function After Interscalene Brachial Plexus Block: a Dose-finding Study
Brief Title: The Minimum Effective Dose (ED90) of Liposomal Bupivacaine for Preserving Motor Function
Acronym: ED90
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, Dr., Affiliated Hospital of Jiaxing University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2024-KY-656-002
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Motion Sickness
Keywords: Shoulder surgery; Intermuscular sulcus brachial plexus block; Bupivacaine liposome; Effective dose
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First patient's dose of bupivacaine liposome (Experimental): First patient's use of bupivacaine liposome and next patient's use of bupivacaine liposome
  Interventions: Drug: First patient Bupivacaine liposome and next patient Bupivacaine liposome
- next patient's dose of bupivacaine liposome (Experimental): First patient's use of bupivacaine liposome and next patient's use of bupivacaine liposome
  Interventions: Drug: First patient Bupivacaine liposome and next patient Bupivacaine liposome

INTERVENTIONS:
Drug: First patient Bupivacaine liposome and next patient Bupivacaine liposome — This study was conducted using the biased coin method, where each patient's use of bupivacaine liposome dose depended on the previous patient's response. Based on previous research and our past experience, the first recruited patient used a dose of 66.5mg (15ml). Subsequently, if motor function was preserved, the next patient received a higher dose (increased by 6.65mg) with a probability of b=0.11; or the same dose with a probability of 1-b=0.89. If motor function was blocked, the next patient received a lower dose (decreased by 6.65mg).

SUMMARY:
Explore the minimum effective dose of liposomal bupivacaine for preserving motor function

DETAILED DESCRIPTION:
Our research group plans to conduct a dose exploration experiment, using a biased coin design sequential method to explore the 90% minimum effective dose of bupivacaine liposomes for preserving motor function after intermuscular groove brachial plexus block surgery in shoulder arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

Age 41-65 years ASA physical condition 1-3 BMI 18-30 kg/m2 undergoing arthroscopic shoulder surgery

Exclusion Criteria:

Inability to consent to the study pregnancy allergy to local anesthetics preexisting neuropathy cervical pathologies (i.e., herniated disc, myelopathy) chronic pain syndromes (defined as reflex sympathetic dystrophy or complex regional pain syndrome) severe respiratory conditions psychiatric or cognitive disorders that prohibit patients from adhering to the study protocol history of drug or alcohol abuse chronic opioid use (longer than 3 months or daily morphine equivalents more than 5mg/day for 1 month) contraindication for general anesthesia and/or interscalene nerve block and planned open shoulder arthrotomies Muscle related diseases

Ages: 41 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
ED90 of motor function was preserved 72 hours after brachial plexus block | 72 hours after brachial plexus block
  Evaluate the effective sensory blockade for maintaining motor function at the time point

CONTACTS AND LOCATIONS:
Overall Officials: Qinghe Zhou, Study Chair — Affiliated Hospital of Jiaxing University
Locations (1):
- Affiliated Hospital of Jiaxing University, Jiaxing, China

IPD SHARING:
Plan to Share IPD: No